CLINICAL TRIAL: NCT04192292
Title: Study of Sulphonylurea Synergy With DPP4 Inhibitors
Acronym: SSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018DM13
Record Dates: First submitted 2019-10-09; First posted 2019-12-10 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes
Keywords: Metformin; Sulphonylurea; Gliclazide; DPP4 Inhibitor; Sitagliptin; Continuous Glucose Monitoring; KCNJ11; Incretin Effect
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sulfonylurea Compounds; Gliclazide; Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Intervention Model Description: Physiological Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Treatment (No Intervention): No change to participants standard care
- Low dose sulphonylurea alone (Experimental): Participants will be given a single dose of low dose sulphonylurea once daily for 14 days as a physiological stimulus. The sulphonylurea given in this study will be gliclazide 20mg orally once daily.
  Interventions: Drug: Sulfonylurea
- DPP4 inhibitor alone (Experimental): Participants will be given a single dose of DPP4 inhibitor once daily for 14 days as a physiological stimulus. The DPP inhibitor given in this study will be sitagliption 100mg orally once daily.
  Interventions: Drug: DPP4 Inhibitor
- Low dose sulphonylurea + DPP4 inhibitor (Experimental): Participants will be given a single dose of low dose sulphonylurea once daily and a single dose of DPP4 inhibitor for 14 days as a physiological stimulus. The sulphonylurea given in this study will be gliclazide 20mg orally once daily and the DPP4 inhibitor will be sitagliptin orally100mg once daily.
  Interventions: Drug: Sulfonylurea; Drug: DPP4 Inhibitor

INTERVENTIONS:
Drug: Sulfonylurea — Given at very low dose as a physiological stimulus on the beta cell not as medical treatment. 20mg gliclazide is being used in this study.
  Other Names: Diamicron; Nordialex; Gliclazide
  Arms: Low dose sulphonylurea + DPP4 inhibitor; Low dose sulphonylurea alone
Drug: DPP4 Inhibitor — Given as a physiological stimulus to augment endogenous incretin hormone levels, not as a medical treatment. 100mg sitagliptin is being used in this study.
  Other Names: Sitagliptin; Januvia; Janumet; Ristaben; Tesavel; Velmetia; Xelevia
  Arms: DPP4 inhibitor alone; Low dose sulphonylurea + DPP4 inhibitor

SUMMARY:
The Study of Sulphonylurea Synergy with DPP4 Inhibitors (SSS Study) will establish whether a very low dose of sulphonylurea will have a synergistic role on augmentation of insulin secretion when given in combination with a DPP4 inhibitor as a primary outcome. The study will recruit 30 patients with type 2 diabetes mellitus controlled with no treatment or metformin monotherapy with an HbA1c <64mmol/mol (<8%). In this unblinded, randomised physiological study, participants will receive four 14-day intervention blocks: low dose sulphonylurea alone, DPP4 inhibitor alone, low dose sulphonylurea + DPP4 inhibitor or no treatment change. The primary outcome will be assessed through evaulation of insulin secretion and sensitivity at mixed meal test at the end of each treatment block. Glycaemic variability on continuous glucose monitoring for each intervention block will be evaluated as a secondary outcome. In addition, the primary outcome will be evaulated for KCNJ11 genotype as an additional secondary outcome.

DETAILED DESCRIPTION:
The Study of Sulphonylurea Synergy with DPP4 Inhibitors (SSS Study) aims to establish whether a very low dose of SU will have a synergistic role to increase insulin secretion when given in combination with DPP4 inhibitors (DPP4i). This physiological study will assess glucose variability and insulin secretion through mixed meal tests and continuous glucose monitoring.

The SSS Study is a follow-on study from The Study of Sulphonylurea Synergy with Incretins (LOGIC Study 2018DM01, 18/ES/0064, ClinicalTrials.gov NCT03705195) which established that the use of low dose sulphonylurea as a physiological stimulus augments insulin secretion through synergistic action with incretin hormones.

In this study, low dose sulphonylurea will again be used as a physiological stimulus. A DPP4i will be given to increase levels of incretin hormones. The investigator's hypothesis is that a combination of low-dose sulphonylurea with a DPP4i will further augment insulin secretion than with low-dose SU alone. In addition, utilising results from LOGIC Study, the low-dose SU has been shown to promote insulin secretion in a glucose-dependent mechanism via synergy with incretin hormones, therefore glycaemic variability should be minimised.

The SSS study will take place at The Clinical Research Centre in Dundee over 6 visits. It will evaluate 30 patients with T2DM on no diabetes therapy or metformin monotherapy. All participants will continue their existing diabetes treatment for the duration of the study.

SSS Study clinical stage will be 8 weeks. A screening visit will obtain Informed Written Consent for Study, along with baseline medical information and screening bloods to ensure the participant is safe to take part.

There are four, 2-week blocks during the clinical phase of the study:

* Block 1: No change to treatment
* Block 2: Low Dose Sulphonylurea Once Daily
* Block 3: DPP4i Once Daily
* Block 4: Low Dose Sulphonylurea + DPP4i Once Daily

The SSS Study is randomised to intervention order. Participants will crossover to receive each intervention during the study period. They will be randomised using a computer randomisation software.

At the four intensive visits, participants will undergo a two-hour MMT to assess post-prandial glucose variance. In addition, participants will wear CGM (Freestyle Libre Pro Flash Continuous Glucose Monitoring System, Abbot) for the duration of study to assess overall physiological glucose variability. The CGM sensor will be replaced at each study visit. The CGM has a dedicated software, meters will be downloaded to a secure University computer. The software produces an analysis of blood sugar readings for the last 14 days.

Comparison of glycaemic variability and post-prandial insulin secretion after each of the treatment periods will investigate whether low-dose SU and DPP4i further augment insulin secretion compared with low-dose SU alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧40 and ≦80
* Age of diabetes diagnosis ≧35
* T2DM on no treatment, or metformin monotherapy
* White British
* HbA1c ≦8% (64mmol/mol) in last 6 months
* eGFR ≧50ml/min-1
* ALT ≦2.5*ULN
* Able to consent

Exclusion Criteria:

* Does not meet inclusion criteria
* Pregnancy, lactation or a female planning to conceive within the study period
* Previous acute pancreatitis
* Established pancreatic disease
* Participating in clinical phase of another interventional trial/study or have done so within the last 30 days.
* Any other significant medical reason for exclusion as determined by the investigator
* Inability or unwillingness to comply with protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Difference in incretin effect between mixed meal tests | Through four mixed meal tests which take place at the end of each 14 day intervention block. The four intervention blocks will be completed during an 8 week clinical phase of study.
  Comparison of four mixed meal tests performed at the end of each intervention block. Meal tests will evaluate 1) No intervention 2) Low dose sulphonylurea alone 3) DPP4 inhibitor alone 4) Low dose sulphonylurea + DPP4 inhibitor. Measures of the incretin effect will be compared between the different blocks.

SECONDARY OUTCOMES:
Insulin secretory response analysed by KCNJ11 genotype | Through 4 meal test visits completed over an 8 week clinical phase of study. Outcome will also be evaluated through variability of glucose levels observed on continuous glucose monitoring worn for duration of 8 week clinical phase.
  Difference in insulin secretory response to low dose gliclazide calculated by insulin/cpeptide levels in each meal test visit. Differences will then be compared by participants genotype e.g. insulin secretory response for E23K, E23E, K23K variants.
Variation in blood glucose during intervention blocks analysed by continuous glucose monitoring | Meansurements taken via continuous glucose monitoring sensors worn by participants for duration of 8 week clinical phase
  Comparison time-in-range of blood sugars as low, target and high on continuous glucose monitoring between each intervention block

CONTACTS AND LOCATIONS:
Locations (1):
- Ninewells Hospital and Medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study of Sulphonylurea Synergy with Incretins — https://clinicaltrials.gov/ct2/show/NCT03705195